CLINICAL TRIAL: NCT02678455
Title: Phase II, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Immunogenicity of the Recombinant Live Attenuated Tetravalent Dengue Virus Vaccine Admixture TV005 (TetraVax-DV TV005) in Healthy Adults, Adolescents, and Children in Dhaka, Bangladesh
Brief Title: Safety and Immunogenicity of the Dengue Virus Vaccine TV005 (TetraVax-DV TV005) in Healthy Adults, Adolescents, and Children in Dhaka, Bangladesh
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Vermont (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-15097; Dengue TV005 in Dhaka (Other: NIAID)
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-02

CONDITIONS: Dengue
Keywords: Dengue Virus
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TV005 vaccine (Experimental): Participants will receive one dose of TV005 vaccine at study entry (Day 0).
  Interventions: Biological: TV005 vaccine
- Placebo (Placebo Comparator): Participants will receive one dose of placebo at study entry (Day 0).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TV005 vaccine — Delivered by subcutaneous injection; contains 10^3 PFU of rDEN1Δ30, 10^4 PFU of rDEN2/4Δ30(ME), 10^3 PFU of rDEN3Δ30/31, and 10^3 PFU of rDEN4Δ30.
  Other Names: TetraVax-DV T005
  Arms: TV005 vaccine
Biological: Placebo — Delivered by subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of the recombinant live attenuated tetravalent dengue virus vaccine admixture TV005 (TetraVax-DV T005) in healthy adults, adolescents, and children in Dhaka, Bangladesh.

DETAILED DESCRIPTION:
Dengue viruses (DENV) are the leading arboviral infection globally, with over 2 billion people at risk of infection worldwide. The first dengue fever outbreak in Bangladesh occurred in 2000, and since then, dengue fever has had a continued presence throughout Bangladesh. This study will evaluate the safety and immunogenicity of the recombinant live attenuated tetravalent dengue virus vaccine admixture TV005 (TetraVax-DV T005) in healthy adults, adolescents, and children in Dhaka, Bangladesh.

The study will enroll four cohorts of participants: adults, adolescents, children, and young children. Study researchers will evaluate study data for each cohort before enrolling the subsequent cohort.

Participants will be randomly assigned to receive either TV005 vaccine or placebo at study entry (Day 0). Additional study visits will occur on Days 7, 14, 28, 56, 180, 360, 720, and 1080. Study visits will include blood collection, physical examinations, and clinical assessments. Participants will record and monitor their temperature and symptoms until Day 14. Study staff will contact participants daily until Day 14; after Day 14, study staff will contact participants weekly (and after Day 180, monthly) throughout the study for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females (non-pregnant or lactating) between the ages of 12 months and 50 years at the time of enrollment into the study.
* Reside in Mirpur Wards 2, 3, or 5 (or other Wards within Mirpur as designated by the PI if needed to reach enrollment targets) at the time of screening.
* Study participants and/or their parents/guardians/legally acceptable or authorized representatives (LARs) who the Investigator believes can and will comply with the requirements of the protocol (e.g., return for follow-up visits).
* Good general health as determined by physical examination, laboratory screening, and review of medical history.
* If the participant is greater than or equal to 18 years of age, an informed consent form signed and dated by the study participant (and by an independent witness if required by local regulations). If the study participant is a minor, an assent form (for participants age 11-17 years) and informed consent form signed and dated by the participant's properly identified parent(s) or legally acceptable representative. If a participant is less than 11 years of age, the participant's parent(s) or legally acceptable representative will consent by signing the consent form for minor participants.
* If the participant is female, she must not be pregnant or planning to become pregnant up to 28 days post vaccination. Female participants under the age of 18 will be enrolled, if they have not yet reached menarche. Females 18 years of age or older, must be properly using a method of pregnancy prevention that is known to be highly effective per the PI. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (greater than or equal to 6 months since last sexual encounter). For female study participants who are 18 years of age or older pregnancy testing will occur at screening and again before vaccination and they must have a negative pregnancy test prior to vaccination. Additionally, they will receive counselling on the importance of effective contraception during the 30 days prior to vaccination and continuing up to Day 28. Counselling will occur at their screening visit, on all clinic visit days up to Day 28. Female participants 18 years of age and older will be subject to pregnancy testing on the Study Day 28 and 56 visits. If female participants under the age of 18 that have not yet reached menarche prior to enrollment, reach menarche during the study, they will continue to be enrolled and followed-up through the entire three year follow-up period.

Exclusion Criteria:

* Pregnant or lactating female or female planning to become pregnant within 28 days of receiving an investigational product or planning to discontinue abstinence or contraceptive precautions within 28 days of receiving an investigational product. Menstruating females under the age of 18 will be excluded from being enrolled.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, renal, autoimmune, hematologic, or endocrine disease or functional defect, as determined by history, physical examination, or screening tests.
* History of any neurological, psychiatric, or behavioural disorder or seizures, with the exception of a single febrile seizure in childhood.
* Self-reported or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent, greater than or equal to 0.5 mg/kg/day or 20 mg/day, for more than 2 consecutive weeks within the past 3 months). Inhaled and topical steroids are allowed.
* Having a height-for-age z-score (HAZ) or weight-for-age z-score (WAZ) of less than or equal to 3 for children under the age of two. Severe malnutrition as observed by the study physician for all study participants ages 2 years old and older.
* Hepatitis C virus (HCV) infection by screening and confirmatory assays (screening in adults and adolescents only), or hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening (all participants) or, unwilling to allow HCV (adults and adolescents only) and HBV testing.
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine transaminase (ALT), or platelet count, as defined in this protocol.
* For children under 5 years of age, screening laboratory values of Grade 1 or above for Haemoglobin.
* History of allergic reaction likely to be exacerbated by any component of the vaccine; any history of a severe allergic reaction or anaphylaxis.
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures.
* Any other condition that in the opinion of the Investigator would jeopardize the safety or rights of a participant participating in the trial or would render the participant unable to comply with the protocol.
* Planned administration of any vaccine from 30 days prior to receipt of the study vaccine and ending 30 days after; with the exceptions of standard infant and child Expanded Program on Immunization (EPI) inactivated vaccines and the inactivated influenza vaccine or the inactivated rabies vaccine (without administration of immunoglobulin) administered to adults or children.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding receipt of study vaccine/placebo or planned use at any time during the study period or history of having received any investigational dengue vaccine at any previous time.
* Current participation in any clinical or investigational study.
* Administration of immunoglobulins and/or blood products within 90 days preceding the dose or planned administration at any time during the study period, which might interfere with assessment of the immune response.
* A planned or anticipated move to a location that will prohibit full participation in the trial for the three year duration.
* Potential adult volunteers or parents of potential child volunteers, who do not have easy access to a fixed or mobile telephone.
* Any participant that resides in a household with an individual previously enrolled in an older age cohort in this study. Only one participant from each household will be enrolled.
* Any participant identified as a site employee of the Investigator or study clinic, with direct involvement in the proposed study or other studies under the direction of that Investigator or study clinic, as well as any immediate family member (such as husband, wife and their children, adopted or natural) of the clinic employees or the Investigator.

Elimination Criteria During the Study:

The following criteria should be checked at each visit subsequent to the first visit. If any become applicable during the study, it will not require withdrawal of the participant from the study but may determine a participant's evaluability in the per-protocol (PP) analysis. The participant will continue to be evaluated for safety purposes at the regularly scheduled visits. See the protocol for definition of study cohorts to be evaluated.

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine/placebo during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs during the study period. For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed.
* Administration of a licensed vaccine during the period starting from 30 days before dose of vaccine/placebo and ending 30 days after, with the exception of standard infant and childhood EPI "inactivated" vaccinations.
* Administration of immunoglobulins and/or any blood products during the study period.
* Pregnancy within the 28 days after investigational product administration.

Ages: 12 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 192 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08-10 (Actual); Study Completion 2020-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rashidul Haque, MD, Principal Investigator — Centre for Vaccine Sciences, International Centre for Diarrhoeal Disease Research, Bangladesh; Beth D. Kirkpatrick, MD, Study Chair — Vaccine Testing Center, University of Vermont College of Medicine
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Mīrpur, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Podder G, Breiman RF, Azim T, Thu HM, Velathanthiri N, Mai le Q, Lowry K, Aaskov JG. Origin of dengue type 3 viruses associated with the dengue outbreak in Dhaka, Bangladesh, in 2000 and 2001. Am J Trop Med Hyg. 2006 Feb;74(2):263-5. PMID 16474082
- [Background] Kirkpatrick BD, Durbin AP, Pierce KK, Carmolli MP, Tibery CM, Grier PL, Hynes N, Diehl SA, Elwood D, Jarvis AP, Sabundayo BP, Lyon CE, Larsson CJ, Jo M, Lovchik JM, Luke CJ, Walsh MC, Fraser EA, Subbarao K, Whitehead SS. Robust and Balanced Immune Responses to All 4 Dengue Virus Serotypes Following Administration of a Single Dose of a Live Attenuated Tetravalent Dengue Vaccine to Healthy, Flavivirus-Naive Adults. J Infect Dis. 2015 Sep 1;212(5):702-10. doi: 10.1093/infdis/jiv082. Epub 2015 Mar 22. PMID 25801652
- [Derived] Walsh MR, Alam MS, Pierce KK, Carmolli M, Alam M, Dickson DM, Bak DM, Afreen S, Nazib F, Golam K, Qadri F, Diehl SA, Durbin AP, Whitehead SS, Haque R, Kirkpatrick BD. Safety and durable immunogenicity of the TV005 tetravalent dengue vaccine, across serotypes and age groups, in dengue-endemic Bangladesh: a randomised, controlled trial. Lancet Infect Dis. 2024 Feb;24(2):150-160. doi: 10.1016/S1473-3099(23)00520-0. Epub 2023 Sep 27. PMID 37776876
- See also: International Center for Diarrhoeal Diseases Research, Bangladesh — http://www.icddrb.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TV005 Vaccine | Placebo
Started | 144 | 48
Completed | 135 | 46
Not Completed | 9 | 2

BASELINE CHARACTERISTICS:
Population: Two participants met protocol specified elimination criteria from the non-safety analyses. Analysis of baseline characteristics and Adverse Events are completed on 144 vaccine and 48 placebo recipients. The two participants that met protocol specified elimination criteria were on the vaccine arm and therefore only 142 vaccine and 48 placebo recipients were included in the analyses of proportion seropositive and proportion with recovered vaccine virus and or wild type virus after vaccination
Groups:
- Total: Total of all reporting groups
Arm/Group | TV005 Vaccine | Placebo | Total
Number analyzed (Participants) | 144 | 48 | 192
Age, Customized [Mean (Standard Deviation); unit: Years] — Population: Row population differs from overall because they are subgroups of the overall population. For each of the four subgroups (Adult, Adolescent, Children, and Young children), there are 36 study participants in the TV005 vaccine arm and 12 study participants in the Placebo arm, with a total of 144 in the TV005 vaccine arm and 48 in the Placebo arm.
  Years
    Adult: number analyzed (Participants) | 36 | 12 | 48
    Adult | 32.17 (8.26) | 29.25 (5.10) | 31.44 (8.24)
    Adolescent: number analyzed (Participants) | 36 | 12 | 48
    Adolescent | 12.58 (1.81) | 12.83 (1.64) | 12.65 (1.75)
    Children: number analyzed (Participants) | 36 | 12 | 48
    Children | 8.14 (1.46) | 7.83 (1.34) | 8.06 (1.42)
    Young Children: number analyzed (Participants) | 36 | 12 | 48
    Young Children | 3.25 (0.81) | 3.42 (0.52) | 3.29 (0.74)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Adult Female | 23 | 5 | 28
  Adult Male | 13 | 7 | 20
  Adolescent Female | 17 | 4 | 21
  Adolescent Male | 19 | 8 | 27
  Child Female | 26 | 7 | 33
  Child Male | 10 | 5 | 15
  Young Child Female | 14 | 5 | 19
  Young Child Male | 22 | 7 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 144 | 48 | 192
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Bangladesh | 144 | 48 | 192
Dengue Serostatus [Count of Participants; unit: Participants]
  Dengue Naive | 81 | 22 | 103
  Dengue Experienced | 63 | 26 | 89
Age Cohort [Count of Participants; unit: Participants]
  Adult group (18-50 years) | 36 | 12 | 48
  Adolescent group (11-17 years) | 36 | 12 | 48
  Children group (5-10 years) | 36 | 12 | 48
  Young children group (1-4 years) | 36 | 12 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Study Participants With Each Solicited, Related Adverse Event Types of Any Severity.
Description: Collected through daily home visits up to day 14, clinic visits for physical exam and hematological and blood chemistry labs, and weekly phone surveillance after day 14. Study staff record temperatures and AEs on the surveillance source document.
Time Frame: Vaccine/placebo administration (study day 0) up to 28 days post vaccine/placebo administration
Population: Per Protocol: all participants who received study vaccine/placebo according to random assignment according to dose are in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TV005 Vaccine | Placebo
Number analyzed (Participants) | 144 | 48
Participants
  Erythema | 1 | 0
  Swelling | 1 | 0
  ALT Increased | 5 | 2
  Hemoglobin Decreased | 5 | 2
  Leukocytosis | 2 | 1
  PTT Prolonged | 4 | 2
  Thrombocytopenia | 4 | 0
  Fever | 7 | 0
  Headache | 17 | 7
  Rash | 37 | 6
  Arthralgia | 7 | 0
  Fatigue | 7 | 2
  Myalgia | 7 | 1
  Nausea | 6 | 2
  Photophobia | 1 | 0
  Retro-orbital Pain | 3 | 1
  Decrease in Activity | 1 | 0
  Loss of Appetite | 1 | 0
  Vomiting | 3 | 0
Statistical Analysis 1: Comparison: TV005 Vaccine vs Placebo; Erythema; Test type: Superiority; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.216 to 0.141] — Adjusted proportion difference (TV005 minus Placebo) with inverse variance weighting and Newcombe Score confidence intervals
Statistical Analysis 2: Comparison: TV005 Vaccine vs Placebo; Swelling; Test type: Superiority; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.216 to 0.141] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: TV005 Vaccine vs Placebo; ALT Increased; Test type: Superiority; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.135 to 0.119] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: TV005 Vaccine vs Placebo; Hemoglobin Decreased; Test type: Superiority; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.135 to 0.119] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: TV005 Vaccine vs Placebo; Leukocytosis; Test type: Superiority; Risk Difference (RD) = 0.020, 95% CI 2-sided [-0.205 to 0.121] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: TV005 Vaccine vs Placebo; PTT Prolonged; Test type: Superiority; Risk Difference (RD) = 0.024, 95% CI 2-sided [-0.127 to 0.111] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: TV005 Vaccine vs Placebo; Thrombocytopenia; Test type: Superiority; Risk Difference (RD) = 0.056, 95% CI 2-sided [0.022 to 0.134] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: TV005 Vaccine vs Placebo; Fever; Test type: Superiority; Risk Difference (RD) = 0.051, 95% CI 2-sided [0.018 to 0.118] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: TV005 Vaccine vs Placebo; Headache; Test type: Superiority; Risk Difference (RD) = -0.036, 95% CI 2-sided [-0.203 to 0.089] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: TV005 Vaccine vs Placebo; Rash; Test type: Superiority; Risk Difference (RD) = 0.166, 95% CI 2-sided [0.016 to 0.275] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: TV005 Vaccine vs Placebo; Arthralgia; Test type: Superiority; Risk Difference (RD) = 0.063, 95% CI 2-sided [0.030 to 0.126] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: TV005 Vaccine vs Placebo; Fatigue; Test type: Superiority; Risk Difference (RD) = 0.023, 95% CI 2-sided [-0.155 to 0.118] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: TV005 Vaccine vs Placebo; Myalgia; Test type: Superiority; Risk Difference (RD) = 0.041, 95% CI 2-sided [-0.105 to 0.105] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: TV005 Vaccine vs Placebo; Nausea; Test type: Superiority; Risk Difference (RD) = 0.019, 95% CI 2-sided [-0.160 to 0.114] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: TV005 Vaccine vs Placebo; Photophobia; Test type: Superiority; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.216 to 0.141] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: TV005 Vaccine vs Placebo; Retro-orbital Pain; Test type: Superiority; Risk Difference (RD) = 0.024, 95% CI 2-sided [-0.142 to 0.088] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: TV005 Vaccine vs Placebo; Decrease in Activity; Test type: Superiority; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.216 to 0.141] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: TV005 Vaccine vs Placebo; Loss of Appetite; Test type: Superiority; Risk Difference (RD) = 0.028, 95% CI 2-sided [-0.216 to 0.141] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: TV005 Vaccine vs Placebo; Vomiting; Test type: Superiority; Risk Difference (RD) = 0.083, 95% CI 2-sided [-0.165 to 0.218] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Study Participants Who Are Seropositive Following Vaccination
Description: Measured by serum plaque reduction neutralization titer, 50% (PRNT50) to DENV-1, DENV-2, DENV-3, and DENV-4 viruses at study day 14, 28, 58, and 180 post vaccination. Seropositivity to each serotype as defined as PRNT50>=10.
  Per protocol analysis includes participants meeting eligibility criteria, complying with defined visits and protocols, no elimination criteria, and immunogenicity data endpoints measures available.
Time Frame: Study day 14 through study day 180
Population: Only TV005 Vaccine arm included in analysis as per protocol to determine percentage of participants in TV005 vaccine arm who are seropositive after vaccination. Data is analyzed for each sub-group. Two participants (one each in Adult and Adolescent vaccine group) were eliminated from this analysis. There are 35 participants in Adult and Adolescent vaccine Arm groups; 36 in Children, and Young Children vaccine Arm groups with a total of 142 included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TV005 Vaccine
Number analyzed (Participants) | 142
Percentage of participants
  All study participants seropositive to DENV-1 post TV005 Vaccination | 83 [76 to 88]
  All study participants seropositive to DENV-2 post TV005 Vaccination | 99 [96 to 100]
  All study participants seropositive to DENV-3 post TV005 Vaccination | 96 [92 to 98]
  All study participants seropositive to DENV-4 post TV005 Vaccination | 87 [81 to 92]
  Adult study participants seropositive to DENV-1 post TV005 vaccination: number analyzed (Participants) | 35
  Adult study participants seropositive to DENV-1 post TV005 vaccination | 86 [71 to 94]
  Adult study participants seropositive to DENV-2 post TV005 vaccination: number analyzed (Participants) | 35
  Adult study participants seropositive to DENV-2 post TV005 vaccination | 97 [85 to 99]
  Adult study participants seropositive to DENV-3 post TV005 vaccination: number analyzed (Participants) | 35
  Adult study participants seropositive to DENV-3 post TV005 vaccination | 97 [85 to 99]
  Adult study participants seropositive to DENV-4 post TV005 vaccination: number analyzed (Participants) | 35
  Adult study participants seropositive to DENV-4 post TV005 vaccination | 91 [78 to 97]
  Adolescent study participants seropositive to DENV-1 post TV005 vaccination: number analyzed (Participants) | 35
  Adolescent study participants seropositive to DENV-1 post TV005 vaccination | 83 [67 to 92]
  Adolescent study participants seropositive to DENV-2 post TV005 vaccination: number analyzed (Participants) | 35
  Adolescent study participants seropositive to DENV-2 post TV005 vaccination | 100 [90 to 100]
  Adolescent study participants seropositive to DENV-3 post TV005 vaccination: number analyzed (Participants) | 35
  Adolescent study participants seropositive to DENV-3 post TV005 vaccination | 97 [85 to 99]
  Adolescent study participants seropositive to DENV-4 post TV005 vaccination: number analyzed (Participants) | 35
  Adolescent study participants seropositive to DENV-4 post TV005 vaccination | 86 [71 to 94]
  Children study participants seropositive to DENV-1 post TV005 vaccination: number analyzed (Participants) | 36
  Children study participants seropositive to DENV-1 post TV005 vaccination | 81 [65 to 90]
  Children study participants seropositive to DENV-2 post TV005 vaccination: number analyzed (Participants) | 36
  Children study participants seropositive to DENV-2 post TV005 vaccination | 100 [90 to 100]
  Children study participants seropositive to DENV-3 post TV005 vaccination: number analyzed (Participants) | 36
  Children study participants seropositive to DENV-3 post TV005 vaccination | 100 [90 to 100]
  Children study participants seropositive to DENV-4 post TV005 vaccination: number analyzed (Participants) | 36
  Children study participants seropositive to DENV-4 post TV005 vaccination | 78 [62 to 88]
  Young children study participants seropositive to DENV-1 post TV005 vaccination: number analyzed (Participants) | 36
  Young children study participants seropositive to DENV-1 post TV005 vaccination | 83 [68 to 92]
  Young children study participants seropositive to DENV-2 post TV005 vaccination: number analyzed (Participants) | 36
  Young children study participants seropositive to DENV-2 post TV005 vaccination | 100 [90 to 100]
  Young children study participants seropositive to DENV-3 post TV005 vaccination: number analyzed (Participants) | 36
  Young children study participants seropositive to DENV-3 post TV005 vaccination | 92 [78 to 97]
  Young children study participants seropositive to DENV-4 post TV005 vaccination: number analyzed (Participants) | 36
  Young children study participants seropositive to DENV-4 post TV005 vaccination | 94 [82 to 98]
Statistical Analysis 1: Comparison: TV005 Vaccine; All study participants seropositive to DENV-1 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 83, 95% CI 2-sided [76 to 88]
Statistical Analysis 2: Comparison: TV005 Vaccine; All study participants seropositive to DENV-2 post TV005 Vaccination. There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 99, 95% CI 2-sided [96 to 100]
Statistical Analysis 3: Comparison: TV005 Vaccine; All study participants seropositive to DENV-3 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 96, 95% CI 2-sided [92 to 98]
Statistical Analysis 4: Comparison: TV005 Vaccine; All study participants seropositive to DENV-4 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 87, 95% CI 2-sided [81 to 92]
Statistical Analysis 5: Comparison: TV005 Vaccine; Adult study participants seropositive to DENV-1 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 86, 95% CI 2-sided [71 to 94]
Statistical Analysis 6: Comparison: TV005 Vaccine; Adult study participants seropositive to DENV-2 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 97, 95% CI 2-sided [85 to 99]
Statistical Analysis 7: Comparison: TV005 Vaccine; Adult study participants seropositive to DENV-3 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 97, 95% CI 2-sided [85 to 99]
Statistical Analysis 8: Comparison: TV005 Vaccine; Adult study participants seropositive to DENV-4 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 91, 95% CI 2-sided [78 to 97]
Statistical Analysis 9: Comparison: TV005 Vaccine; Adolescent study participants seropositive to DENV-1 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 83, 95% CI 2-sided [67 to 92]
Statistical Analysis 10: Comparison: TV005 Vaccine; Adolescent study participants seropositive to DENV-2 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 100, 95% CI 2-sided [90 to 100]
Statistical Analysis 11: Comparison: TV005 Vaccine; Adolescent study participants seropositive to DENV-3 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 97, 95% CI 2-sided [85 to 99]
Statistical Analysis 12: Comparison: TV005 Vaccine; Adolescent study participants seropositive to DENV-4 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 86, 95% CI 2-sided [71 to 94]
Statistical Analysis 13: Comparison: TV005 Vaccine; Children study participants seropositive to DENV-1 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 81, 95% CI 2-sided [65 to 90]
Statistical Analysis 14: Comparison: TV005 Vaccine; Children study participants seropositive to DENV-2 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 100, 95% CI 2-sided [90 to 100]
Statistical Analysis 15: Comparison: TV005 Vaccine; Children study participants seropositive to DENV-3 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 100, 95% CI 2-sided [90 to 100]
Statistical Analysis 16: Comparison: TV005 Vaccine; Children study participants seropositive to DENV-4 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 78, 95% CI 2-sided [62 to 88]
Statistical Analysis 17: Comparison: TV005 Vaccine; Young Children study participants seropositive to DENV-1 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 83, 95% CI 2-sided [68 to 92]
Statistical Analysis 18: Comparison: TV005 Vaccine; Young Children study participants seropositive to DENV-2 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 100, 95% CI 2-sided [90 to 100]
Statistical Analysis 19: Comparison: TV005 Vaccine; Young Children study participants seropositive to DENV-3 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 92, 95% CI 2-sided [78 to 97]
Statistical Analysis 20: Comparison: TV005 Vaccine; Young Children study participants seropositive to DENV-4 post TV005 Vaccination There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 94, 95% CI 2-sided [82 to 98]

3. Secondary Outcome: Proportion of Study Participants With Vaccine Virus Recovered Following Vaccination
Description: Viremia in serum was determined both by amplification and direct titration using Vero cell monolayers. Each specific serotype was identified using monoclonal antibodies.
Time Frame: Vaccine administration (study day 0) up to 14 days post vaccine administration
Population: Per protocol analysis includes all study participants meeting all eligibility criteria and with viremia data endpoints measures available.
Measure: Count of Participants; unit: Participants
Arm/Group | TV005 Vaccine | Placebo
Number analyzed (Participants) | 142 | 48
Participants
  DENV-1 recovered | 4 | 0
  DENV-2 recovered | 1 | 0
  DENV-3 recovered | 1 | 0
  DENV-4 recovered | 0 | 0
  Total Viremia recovered | 6 | 0

4. Secondary Outcome: Percentage of Seropositive Study Participants Among Dengue Experienced and Dengue Naive Vaccinees.
Description: Measured by serum plaque reduction neutralization titer, 50% (PRNT50) to DENV-1, DENV-2, DENV-3, and DENV-4 viruses at study day 14, 28, 56, and 180 post vaccination. Seropositivity to each serotype is defined as PRNT50 ≥ 10.
Time Frame: Study day 14 through study day 180
Population: Only TV005 Vaccine arm included in analysis as per protocol to determine percentage of participants in TV005 vaccine arm who are seropositive after vaccination. Data is analyzed by sub-groups based on previous exposure to Dengue at baseline (experienced, and naïve). Two participants from the experienced at baseline group were eliminated from this analysis. There are 61 participants in the experienced at baseline group; 81 in the naïve at baseline group; total of 142 included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TV005 Vaccine
Number analyzed (Participants) | 142
Percentage of participants
  Experienced at baseline serpositive to DENV-1 post TV005 vaccination: number analyzed (Participants) | 61
  Experienced at baseline serpositive to DENV-1 post TV005 vaccination | 100 [94 to 100]
  Experienced at baseline seropositive to DENV-2 post TV005 vaccination: number analyzed (Participants) | 61
  Experienced at baseline seropositive to DENV-2 post TV005 vaccination | 100 [94 to 100]
  Experienced at baseline seropositive to DENV-3 post TV005 vaccination: number analyzed (Participants) | 61
  Experienced at baseline seropositive to DENV-3 post TV005 vaccination | 100 [94 to 100]
  Experienced at baseline seropoisitive to DENV-4 post TV005 vaccination: number analyzed (Participants) | 61
  Experienced at baseline seropoisitive to DENV-4 post TV005 vaccination | 87 [76 to 93]
  Naive at baseline seropositive to DENV-1 post TV005 vaccination: number analyzed (Participants) | 81
  Naive at baseline seropositive to DENV-1 post TV005 vaccination | 70 [60 to 79]
  Naive at baseline seropositive to DENV-2 post TV005 vaccination: number analyzed (Participants) | 81
  Naive at baseline seropositive to DENV-2 post TV005 vaccination | 99 [93 to 100]
  Naive at baseline seropositive to DENV-3 post TV005 vaccination: number analyzed (Participants) | 81
  Naive at baseline seropositive to DENV-3 post TV005 vaccination | 94 [86 to 97]
  Naive at baseline seropositive to DENV-4 post TV005 vaccination: number analyzed (Participants) | 81
  Naive at baseline seropositive to DENV-4 post TV005 vaccination | 88 [79 to 93]
Statistical Analysis 1: Comparison: TV005 Vaccine; DENV-1 percent seropositive post TV005 vaccination: difference between experienced at baseline and naive at baseline; Test type: Superiority; p < 0.001, Fisher Exact — Comparison between experienced vs dengue naive volunteers post TV005 vaccination. Logistic model to adjust for age cohort provides unstable estimates due to quasi separation of data
Statistical Analysis 2: Comparison: TV005 Vaccine; DENV-2 percent seropositive post TV005 vaccination: difference between experienced at baseline and naive at baseline; Test type: Superiority; p = 1.00, Fisher Exact — Comparison between experienced vs. dengue naive volunteers post TV005 vaccination. Logistic model to adjust for age cohort provides unstable estimates due to quasi separation of data
Statistical Analysis 3: Comparison: TV005 Vaccine; DENV-3 percent seropositive post TV005 vaccination: difference between experienced at baseline and naive at baseline; Test type: Superiority; p = 0.070, Fisher Exact — [p-value comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: TV005 Vaccine; DENV-4 percent seropositive post TV005 vaccination: difference between experienced at baseline and naive at baseline; Test type: Superiority; p = 1.00, Fisher Exact — [p-value comment as in outcome 4, analysis 2]

5. Secondary Outcome: Durability of Seropositivity Post TV005 Vaccination
Description: Estimated percent seropositive, over 3 years by age group and serotype. Measured by serum plaque reduction neutralization titer, 50% (PRNT50) to DENV-1, DENV-2, DENV-3, and DENV-4 viruses at study day 14, 28, 56, 180, 360, 720, and 1080 post vaccination. Seropositivity to each serotype is defined as PRNT50 ≥ 10.
Time Frame: Vaccine/placebo administration (study day 0) up to three years post vaccine/placebo administration (study day 1080).
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TV005 Vaccine
Number analyzed (Participants) | 142
percentage of participants
  Adult cohort: percent seropositive to DENV-1 at study day 0: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-1 at study day 0 | 66 [49 to 79]
  Adult cohort: percent seropositive to DENV-1 at study day 28: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-1 at study day 28 | 83 [67 to 92]
  Adult cohort: percent seropositive to DENV-1 at study day 56: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-1 at study day 56 | 80 [64 to 90]
  Adult cohort: percent seropositive to DENV-1 at study day 180: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-1 at study day 180 | 80 [64 to 90]
  Adult cohort: percent seropositive to DENV-1 at study day 360: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-1 at study day 360 | 80 [64 to 90]
  Adult cohort: percent seropositive to DENV-1 at study day 720: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-1 at study day 720 | 66 [49 to 79]
  Adult cohort: percent seropositive to DENV-1 at study day 1080: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-1 at study day 1080 | 66 [49 to 79]
  Adult cohort: percent seropositive to DENV-2 at study day 0: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-2 at study day 0 | 69 [52 to 81]
  Adult cohort: percent seropositive to DENV-2 at study day 28: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-2 at study day 28 | 94 [81 to 98]
  Adult cohort: percent seropositive to DENV-2 at study day 56: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-2 at study day 56 | 97 [85 to 99]
  Adult cohort: percent seropositive to DENV-2 at study day 180: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-2 at study day 180 | 89 [74 to 95]
  Adult cohort: percent seropositive to DENV-2 at study day 360: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-2 at study day 360 | 89 [74 to 95]
  Adult cohort: percent seropositive to DENV-2 at study day 720: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-2 at study day 720 | 91 [78 to 97]
  Adult cohort: percent seropositive to DENV-2 at study day 1080: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-2 at study day 1080 | 86 [71 to 94]
  Adult cohort: percent seropositive to DENV-3 at study day 0: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-3 at study day 0 | 71 [55 to 84]
  Adult cohort: percent seropositive to DENV-3 at study day 28: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-3 at study day 28 | 94 [81 to 98]
  Adult cohort: percent seropositive to DENV-3 at study day 56: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-3 at study day 56 | 91 [78 to 97]
  Adult cohort: percent seropositive to DENV-3 at study day 180: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-3 at study day 180 | 89 [74 to 95]
  Adult cohort: percent seropositive to DENV-3 at study day 360: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-3 at study day 360 | 86 [71 to 94]
  Adult cohort: percent seropositive to DENV-3 at study day 720: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-3 at study day 720 | 89 [74 to 95]
  Adult cohort: percent seropositive to DENV-3 at study day 1080: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-3 at study day 1080 | 80 [64 to 90]
  Adult cohort: percent seropositive to DENV-4 at study day 0: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-4 at study day 0 | 20 [10 to 36]
  Adult cohort: percent seropositive to DENV-4 at study day 28: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-4 at study day 28 | 77 [61 to 88]
  Adult cohort: percent seropositive to DENV-4 at study day 56: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-4 at study day 56 | 80 [64 to 90]
  Adult cohort: percent seropositive to DENV-4 at study day 180: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-4 at study day 180 | 74 [58 to 86]
  Adult cohort: percent seropositive to DENV-4 at study day 360: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-4 at study day 360 | 66 [49 to 79]
  Adult cohort: percent seropositive to DENV-4 at study day 720: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-4 at study day 720 | 60 [44 to 74]
  Adult cohort: percent seropositive to DENV-4 at study day 1080: number analyzed (Participants) | 35
  Adult cohort: percent seropositive to DENV-4 at study day 1080 | 63 [46 to 77]
  Adolescent cohort: percent seropositive to DENV-1 at study day 0: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-1 at study day 0 | 26 [14 to 42]
  Adolescent cohort: percent seropositive to DENV-1 at study day 28: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-1 at study day 28 | 74 [58 to 86]
  Adolescent cohort: percent seropositive to DENV-1 at study day 56: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-1 at study day 56 | 71 [55 to 84]
  Adolescent cohort: percent seropositive to DENV-1 at study day 180: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-1 at study day 180 | 71 [55 to 84]
  Adolescent cohort: percent seropositive to DENV-1 at study day 360: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-1 at study day 360 | 69 [52 to 81]
  Adolescent cohort: percent seropositive to DENV-1 at study day 720: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-1 at study day 720 | 43 [28 to 59]
  Adolescent cohort: percent seropositive to DENV-1 at study day 1080: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-1 at study day 1080 | 46 [30 to 62]
  Adolescent cohort: percent seropositive to DENV-2 at study day 0: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-2 at study day 0 | 34 [21 to 51]
  Adolescent cohort: percent seropositive to DENV-2 at study day 28: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-2 at study day 28 | 100 [90 to 100]
  Adolescent cohort: percent seropositive to DENV-2 at study day 56: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-2 at study day 56 | 97 [85 to 99]
  Adolescent cohort: percent seropositive to DENV-2 at study day 180: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-2 at study day 180 | 97 [85 to 99]
  Adolescent cohort: percent seropositive to DENV-2 at study day 360: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-2 at study day 360 | 85 [71 to 94]
  Adolescent cohort: percent seropositive to DENV-2 at study day 720: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-2 at study day 720 | 74 [58 to 86]
  Adolescent cohort: percent seropositive to DENV-2 at study day 1080: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-2 at study day 1080 | 69 [52 to 81]
  Adolescent cohort: percent seropositive to DENV-3 at study day 0: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-3 at study day 0 | 37 [23 to 54]
  Adolescent cohort: percent seropositive to DENV-3 at study day 28: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-3 at study day 28 | 89 [74 to 95]
  Adolescent cohort: percent seropositive to DENV-3 at study day 56: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-3 at study day 56 | 94 [81 to 98]
  Adolescent cohort: percent seropositive to DENV-3 at study day 180: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-3 at study day 180 | 97 [85 to 99]
  Adolescent cohort: percent seropositive to DENV-3 at study day 360: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-3 at study day 360 | 89 [74 to 95]
  Adolescent cohort: percent seropositive to DENV-3 at study day 720: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-3 at study day 720 | 57 [41 to 72]
  Adolescent cohort: percent seropositive to DENV-3 at study day 1080: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-3 at study day 1080 | 57 [41 to 72]
  Adolescent cohort: percent seropositive to DENV-4 at study day 0: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-4 at study day 0 | 0 [0 to 10]
  Adolescent cohort: percent seropositive to DENV-4 at study day 28: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-4 at study day 28 | 83 [67 to 92]
  Adolescent cohort: percent seropositive to DENV-4 at study day 56: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-4 at study day 56 | 77 [61 to 88]
  Adolescent cohort: percent seropositive to DENV-4 at study day 180: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-4 at study day 180 | 71 [55 to 84]
  Adolescent cohort: percent seropositive to DENV-4 at study day 360: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-4 at study day 360 | 66 [49 to 79]
  Adolescent cohort: percent seropositive to DENV-4 at study day 720: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-4 at study day 720 | 60 [44 to 74]
  Adolescent cohort: percent seropositive to DENV-4 at study day 1080: number analyzed (Participants) | 35
  Adolescent cohort: percent seropositive to DENV-4 at study day 1080 | 43 [28 to 59]
  Children cohort: percent seropositive to DENV-1 at study day 0: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-1 at study day 0 | 31 [18 to 47]
  Children cohort: percent seropositive to DENV-1 at study day 28: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-1 at study day 28 | 69 [53 to 82]
  Children cohort: percent seropositive to DENV-1 at study day 56: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-1 at study day 56 | 61 [45 to 75]
  Children cohort: percent seropositive to DENV-1 at study day 180: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-1 at study day 180 | 56 [40 to 70]
  Children cohort: percent seropositive to DENV-1 at study day 360: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-1 at study day 360 | 42 [27 to 58]
  Children cohort: percent seropositive to DENV-1 at study day 720: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-1 at study day 720 | 42 [27 to 58]
  Children cohort: percent seropositive to DENV-1 at study day 1080: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-1 at study day 1080 | 36 [22 to 54]
  Children cohort: percent seropositive to DENV-2 at study day 0: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-2 at study day 0 | 33 [20 to 50]
  Children cohort: percent seropositive to DENV-2 at study day 28: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-2 at study day 28 | 92 [78 to 97]
  Children cohort: percent seropositive to DENV-2 at study day 56: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-2 at study day 56 | 89 [75 to 96]
  Children cohort: percent seropositive to DENV-2 at study day 180: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-2 at study day 180 | 92 [78 to 97]
  Children cohort: percent seropositive to DENV-2 at study day 360: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-2 at study day 360 | 78 [62 to 88]
  Children cohort: percent seropositive to DENV-2 at study day 720: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-2 at study day 720 | 67 [50 to 80]
  Children cohort: percent seropositive to DENV-2 at study day 1080: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-2 at study day 1080 | 58 [42 to 73]
  Children cohort: percent seropositive to DENV-3 at study day 0: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-3 at study day 0 | 36 [22 to 52]
  Children cohort: percent seropositive to DENV-3 at study day 28: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-3 at study day 28 | 92 [78 to 97]
  Children cohort: percent seropositive to DENV-3 at study day 56: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-3 at study day 56 | 92 [78 to 97]
  Children cohort: percent seropositive to DENV-3 at study day 180: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-3 at study day 180 | 97 [86 to 100]
  Children cohort: percent seropositive to DENV-3 at study day 360: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-3 at study day 360 | 72 [56 to 84]
  Children cohort: percent seropositive to DENV-3 at study day 720: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-3 at study day 720 | 72 [56 to 84]
  Children cohort: percent seropositive to DENV-3 at study day 1080: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-3 at study day 1080 | 67 [50 to 80]
  Children cohort: percent seropositive to DENV-4 at study day 0: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-4 at study day 0 | 11 [4 to 25]
  Children cohort: percent seropositive to DENV-4 at study day 28: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-4 at study day 28 | 72 [56 to 84]
  Children cohort: percent seropositive to DENV-4 at study day 56: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-4 at study day 56 | 56 [40 to 70]
  Children cohort: percent seropositive to DENV-4 at study day 180: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-4 at study day 180 | 44 [30 to 60]
  Children cohort: percent seropositive to DENV-4 at study day 360: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-4 at study day 360 | 28 [16 to 44]
  Children cohort: percent seropositive to DENV-4 at study day 720: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-4 at study day 720 | 25 [14 to 41]
  Children cohort: percent seropositive to DENV-4 at study day 1080: number analyzed (Participants) | 36
  Children cohort: percent seropositive to DENV-4 at study day 1080 | 19 [10 to 35]
  Young Children cohort: percent seropositive to DENV-1 at study day 0: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-1 at study day 0 | 11 [4 to 25]
  Young Children cohort: percent seropositive to DENV-1 at study day 28: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-1 at study day 28 | 78 [62 to 88]
  Young Children cohort: percent seropositive to DENV-1 at study day 56: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-1 at study day 56 | 42 [27 to 58]
  Young Children cohort: percent seropositive to DENV-1 at study day 180: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-1 at study day 180 | 53 [37 to 68]
  Young Children cohort: percent seropositive to DENV-1 at study day 360: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-1 at study day 360 | 28 [16 to 44]
  Young Children cohort: percent seropositive to DENV-1 at study day 720: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-1 at study day 720 | 28 [16 to 44]
  Young Children cohort: percent seropositive to DENV-1 at study day 1080: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-1 at study day 1080 | 28 [16 to 44]
  Young Children cohort: percent seropositive to DENV-2 at study day 0: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-2 at study day 0 | 11 [4 to 25]
  Young Children cohort: percent seropositive to DENV-2 at study day 28: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-2 at study day 28 | 97 [86 to 100]
  Young Children cohort: percent seropositive to DENV-2 at study day 56: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-2 at study day 56 | 86 [71 to 94]
  Young Children cohort: percent seropositive to DENV-2 at study day 180: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-2 at study day 180 | 81 [65 to 90]
  Young Children cohort: percent seropositive to DENV-2 at study day 360: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-2 at study day 360 | 83 [68 to 92]
  Young Children cohort: percent seropositive to DENV-2 at study day 720: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-2 at study day 720 | 72 [56 to 84]
  Young Children cohort: percent seropositive to DENV-2 at study day 1080: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-2 at study day 1080 | 69 [53 to 82]
  Young Children cohort: percent seropositive to DENV-3 at study day 0: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-3 at study day 0 | 8 [3 to 22]
  Young Children cohort: percent seropositive to DENV-3 at study day 28: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-3 at study day 28 | 86 [71 to 94]
  Young Children cohort: percent seropositive to DENV-3 at study day 56: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-3 at study day 56 | 67 [50 to 80]
  Young Children cohort: percent seropositive to DENV-3 at study day 180: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-3 at study day 180 | 50 [34 to 66]
  Young Children cohort: percent seropositive to DENV-3 at study day 360: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-3 at study day 360 | 25 [14 to 41]
  Young Children cohort: percent seropositive to DENV-3 at study day 720: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-3 at study day 720 | 31 [18 to 47]
  Young Children cohort: percent seropositive to DENV-3 at study day 1080: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-3 at study day 1080 | 25 [14 to 41]
  Young Children cohort: percent seropositive to DENV-4 at study day 0: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-4 at study day 0 | 3 [0 to 14]
  Young Children cohort: percent seropositive to DENV-4 at study day 28: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-4 at study day 28 | 89 [75 to 96]
  Young Children cohort: percent seropositive to DENV-4 at study day 56: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-4 at study day 56 | 72 [56 to 96]
  Young Children cohort: percent seropositive to DENV-4 at study day 180: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-4 at study day 180 | 47 [32 to 63]
  Young Children cohort: percent seropositive to DENV-4 at study day 360: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-4 at study day 360 | 28 [16 to 44]
  Young Children cohort: percent seropositive to DENV-4 at study day 720: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-4 at study day 720 | 28 [16 to 44]
  Young Children cohort: percent seropositive to DENV-4 at study day 1080: number analyzed (Participants) | 36
  Young Children cohort: percent seropositive to DENV-4 at study day 1080 | 22 [12 to 38]
Statistical Analysis 1: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-1 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 66, 95% CI 2-sided [49 to 79]
Statistical Analysis 2: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-1 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 83, 95% CI 2-sided [67 to 92]
Statistical Analysis 3: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-1 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 80, 95% CI 2-sided [64 to 90]
Statistical Analysis 4: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-1 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 80, 95% CI 2-sided [64 to 90]
Statistical Analysis 5: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-1 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 80, 95% CI 2-sided [64 to 90]
Statistical Analysis 6: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-1 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 66, 95% CI 2-sided [49 to 79]
Statistical Analysis 7: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-1 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 66, 95% CI 2-sided [49 to 79]
Statistical Analysis 8: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-2 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 69, 95% CI 2-sided [52 to 81]
Statistical Analysis 9: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-2 at stud day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 94, 95% CI 2-sided [81 to 98]
Statistical Analysis 10: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-2 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 97, 95% CI 2-sided [85 to 99]
Statistical Analysis 11: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-2 at study day 180. There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 89, 95% CI 2-sided [74 to 95]
Statistical Analysis 12: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-2 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 89, 95% CI 2-sided [74 to 95]
Statistical Analysis 13: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-2 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 91, 95% CI 2-sided [78 to 97]
Statistical Analysis 14: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-2 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 86, 95% CI 2-sided [71 to 94]
Statistical Analysis 15: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-3 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 71, 95% CI 2-sided [55 to 84]
Statistical Analysis 16: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-3 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 94, 95% CI 2-sided [81 to 98]
Statistical Analysis 17: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-3 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 91, 95% CI 2-sided [78 to 97]
Statistical Analysis 18: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-3 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 89, 95% CI 2-sided [74 to 95]
Statistical Analysis 19: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-3 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 86, 95% CI 2-sided [71 to 94]
Statistical Analysis 20: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-3 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 89, 95% CI 2-sided [74 to 95]
Statistical Analysis 21: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-3 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 80, 95% CI 2-sided [64 to 90]
Statistical Analysis 22: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-4 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 20, 95% CI 2-sided [10 to 36]
Statistical Analysis 23: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-4 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 77, 95% CI 2-sided [61 to 88]
Statistical Analysis 24: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-4 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 80, 95% CI 2-sided [64 to 90]
Statistical Analysis 25: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-4 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 74, 95% CI 2-sided [58 to 86]
Statistical Analysis 26: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-4 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 66, 95% CI 2-sided [49 to 79]
Statistical Analysis 27: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-4 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 60, 95% CI 2-sided [44 to 74]
Statistical Analysis 28: Comparison: TV005 Vaccine; Adult cohort: percent seropositive to DENV-4 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 63, 95% CI 2-sided [46 to 77]
Statistical Analysis 29: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-1 a study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 26, 95% CI 2-sided [14 to 42]
Statistical Analysis 30: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-1 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 74, 95% CI 2-sided [58 to 86]
Statistical Analysis 31: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-1 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 71, 95% CI 2-sided [55 to 84]
Statistical Analysis 32: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-1 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 71, 95% CI 2-sided [55 to 84]
Statistical Analysis 33: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-1 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 69, 95% CI 2-sided [52 to 81]
Statistical Analysis 34: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-1 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 43, 95% CI 2-sided [28 to 59]
Statistical Analysis 35: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-1 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 46, 95% CI 2-sided [30 to 62]
Statistical Analysis 36: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-2 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 34, 95% CI 2-sided [21 to 51]
Statistical Analysis 37: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-2 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 100, 95% CI 2-sided [90 to 100]
Statistical Analysis 38: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-2 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 97, 95% CI 2-sided [85 to 99]
Statistical Analysis 39: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-2 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 97, 95% CI 2-sided [85 to 99]
Statistical Analysis 40: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-2 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 85, 95% CI 2-sided [71 to 94]
Statistical Analysis 41: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-2 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 74, 95% CI 2-sided [58 to 86]
Statistical Analysis 42: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-2 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 69, 95% CI 2-sided [52 to 81]
Statistical Analysis 43: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-3 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 37, 95% CI 2-sided [23 to 54]
Statistical Analysis 44: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-3 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 89, 95% CI 2-sided [74 to 95]
Statistical Analysis 45: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-3 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 94, 95% CI 2-sided [81 to 98]
Statistical Analysis 46: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-3 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 97, 95% CI 2-sided [85 to 99]
Statistical Analysis 47: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-3 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 89, 95% CI 2-sided [74 to 95]
Statistical Analysis 48: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-3 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 57, 95% CI 2-sided [41 to 72]
Statistical Analysis 49: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-3 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 57, 95% CI 2-sided [41 to 72]
Statistical Analysis 50: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-4 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 0, 95% CI 2-sided [0 to 10]
Statistical Analysis 51: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-4 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 83, 95% CI 2-sided [67 to 92]
Statistical Analysis 52: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-4 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 77, 95% CI 2-sided [61 to 88]
Statistical Analysis 53: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-4 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 71, 95% CI 2-sided [55 to 84]
Statistical Analysis 54: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-4 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 66, 95% CI 2-sided [49 to 79]
Statistical Analysis 55: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-4 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 60, 95% CI 2-sided [44 to 74]
Statistical Analysis 56: Comparison: TV005 Vaccine; Adolescent cohort: percent seropositive to DENV-4 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 43, 95% CI 2-sided [28 to 59]
Statistical Analysis 57: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-1 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 31, 95% CI 2-sided [18 to 47]
Statistical Analysis 58: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-1 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 69, 95% CI 2-sided [53 to 82]
Statistical Analysis 59: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-1 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 61, 95% CI 2-sided [45 to 75]
Statistical Analysis 60: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-1 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 56, 95% CI 2-sided [40 to 70]
Statistical Analysis 61: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-1 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 42, 95% CI 2-sided [27 to 58]
Statistical Analysis 62: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-1 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 42, 95% CI 2-sided [27 to 58]
Statistical Analysis 63: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-1 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 36, 95% CI 2-sided [22 to 54]
Statistical Analysis 64: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-2 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 33, 95% CI 2-sided [20 to 50]
Statistical Analysis 65: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-2 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 92, 95% CI 2-sided [78 to 97]
Statistical Analysis 66: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-2 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 89, 95% CI 2-sided [75 to 96]
Statistical Analysis 67: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-2 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 92, 95% CI 2-sided [78 to 97]
Statistical Analysis 68: Comparison: TV005 Vaccine; children cohort: percent seropositive to DENV-2 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 78, 95% CI 2-sided [62 to 88]
Statistical Analysis 69: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-2 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 67, 95% CI 2-sided [50 to 80]
Statistical Analysis 70: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-2 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 58, 95% CI 2-sided [42 to 73]
Statistical Analysis 71: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-3 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 36, 95% CI 2-sided [22 to 52]
Statistical Analysis 72: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-3 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 92, 95% CI 2-sided [78 to 97]
Statistical Analysis 73: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-3 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 92, 95% CI 2-sided [78 to 97]
Statistical Analysis 74: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-3 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 97, 95% CI 2-sided [86 to 100]
Statistical Analysis 75: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-3 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 72, 95% CI 2-sided [56 to 84]
Statistical Analysis 76: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-3 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 72, 95% CI 2-sided [56 to 84]
Statistical Analysis 77: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-3 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 67, 95% CI 2-sided [50 to 80]
Statistical Analysis 78: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-4 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 11, 95% CI 2-sided [4 to 25]
Statistical Analysis 79: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-4 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 72, 95% CI 2-sided [56 to 84]
Statistical Analysis 80: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-4 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 56, 95% CI 2-sided [40 to 70]
Statistical Analysis 81: Comparison: TV005 Vaccine; children cohort: percent seropositive to DENV-4 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 44, 95% CI 2-sided [30 to 60]
Statistical Analysis 82: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-4 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 28, 95% CI 2-sided [16 to 44]
Statistical Analysis 83: Comparison: TV005 Vaccine; Children cohort: percent seropositive to DENV-4 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 25, 95% CI 2-sided [14 to 41]
Statistical Analysis 84: Comparison: TV005 Vaccine; children cohort: percent seropositive to DENV-4 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 19, 95% CI 2-sided [10 to 35]
Statistical Analysis 85: Comparison: TV005 Vaccine; Young children cohort: percent seropositive to DENV-1 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 11, 95% CI 2-sided [4 to 25]
Statistical Analysis 86: Comparison: TV005 Vaccine; Young children cohort: percent seropositive to DENV-1 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 78, 95% CI 2-sided [62 to 88]
Statistical Analysis 87: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-1 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 42, 95% CI 2-sided [27 to 58]
Statistical Analysis 88: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-1 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 53, 95% CI 2-sided [37 to 68]
Statistical Analysis 89: Comparison: TV005 Vaccine; Young children cohort: percent seropositive to DENV-1 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 28, 95% CI 2-sided [16 to 44]
Statistical Analysis 90: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-1 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 28, 95% CI 2-sided [16 to 44]
Statistical Analysis 91: Comparison: TV005 Vaccine; Young children cohort: percent seropositive to DENV-1 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 28, 95% CI 2-sided [16 to 44]
Statistical Analysis 92: Comparison: TV005 Vaccine; Young children cohort: percent seropositive to DENV-2 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 11, 95% CI 2-sided [4 to 25]
Statistical Analysis 93: Comparison: TV005 Vaccine; Young children cohort: percent seropositive to DENV-2 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 97, 95% CI 2-sided [86 to 100]
Statistical Analysis 94: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-2 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 86, 95% CI 2-sided [71 to 94]
Statistical Analysis 95: Comparison: TV005 Vaccine; Young children cohort: percent seropositive to DENV-2 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 81, 95% CI 2-sided [65 to 90]
Statistical Analysis 96: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-2 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 83, 95% CI 2-sided [68 to 92]
Statistical Analysis 97: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-2 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; Slope = 72, 95% CI 2-sided [56 to 84]
Statistical Analysis 98: Comparison: TV005 Vaccine; Young children cohort: percent seropositive to DENV-2 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 69, 95% CI 2-sided [53 to 82]
Statistical Analysis 99: Comparison: TV005 Vaccine; Young children cohort: percent seropositive to DENV-3 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 8, 95% CI 2-sided [3 to 22]
Statistical Analysis 100: Comparison: TV005 Vaccine; Young children cohort: percent seropositive to DENV-3 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 86, 95% CI 2-sided [71 to 94]
Statistical Analysis 101: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-3 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 67, 95% CI 2-sided [50 to 80]
Statistical Analysis 102: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-3 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 50, 95% CI 2-sided [34 to 66]
Statistical Analysis 103: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-3 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 25, 95% CI 2-sided [14 to 41]
Statistical Analysis 104: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-3 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 31, 95% CI 2-sided [18 to 47]
Statistical Analysis 105: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-3 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 25, 95% CI 2-sided [14 to 41]
Statistical Analysis 106: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-4 at study day 0 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 3, 95% CI 2-sided [0 to 14]
Statistical Analysis 107: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-4 at study day 28 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 89, 95% CI 2-sided [75 to 96]
Statistical Analysis 108: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-4 at study day 56 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 72, 95% CI 2-sided [56 to 96]
Statistical Analysis 109: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-4 at study day 180 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 47, 95% CI 2-sided [32 to 63]
Statistical Analysis 110: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-4 at study day 360 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 28, 95% CI 2-sided [16 to 44]
Statistical Analysis 111: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-4 at study day 720 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 28, 95% CI 2-sided [16 to 44]
Statistical Analysis 112: Comparison: TV005 Vaccine; young children cohort: percent seropositive to DENV-4 at study day 1080 There is no comparison between arms. Only the percentage seropositive in the TV005 vaccine arm is being estimated with confidence interval; Test type: Other — Estimate of the percentage in each sub-group in the TV005 vaccine arm; percentage seropositive = 22, 95% CI 2-sided [12 to 38]

ADVERSE EVENTS:
Time Frame: All-cause mortality and SAEs were assessed through three years post-vaccination; solicited and all other adverse events were assessed through 28 days post vaccination
Description: Time frame for solicited adverse events is up to 28 days post vaccination; time frame for SAE and all-cause mortality is three years post vaccination
Arm/Group | TV005 Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/48
Serious Adverse Events (participants affected / at risk) | 6/144 | 0/48
Other Adverse Events (participants affected / at risk) | 95/144 | 25/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TV005 Vaccine (N=144) | Placebo (N=48)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
ALT Increase (Hepatobiliary disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Endocarditis Infective (Cardiac disorders) | 1 (1) | 0 (0)
Typhoid Fever (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TV005 Vaccine (N=144) | Placebo (N=48)
Injection site erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 9 (9) | 4 (4)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 11 (11) | 1 (1)
Headache (General disorders) | 19 (19) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 37 (37) | 6 (6)
Nausea (Gastrointestinal disorders) | 8 (8) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ALT Elevated (Hepatobiliary disorders) | 5 (5) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0)
Retro-orbital pain (Eye disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 8 (8) | 2 (2)
Photophobia (General disorders) | 1 (1) | 0 (0)
Hemoglobin decreasaed (Blood and lymphatic system disorders) | 20 (20) | 9 (9)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
PT Prolonged (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PTT prolonged (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Decreased appetite (General disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT02678455/Prot_SAP_001.pdf
  • Informed Consent Form (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT02678455/ICF_002.pdf